CLINICAL TRIAL: NCT02208440
Title: A Randomized, Two-arm, Prospective, Subject Blind Study to Assess the Safety and Efficacy of InSpace™ Device in Comparison to Full Thickness Massive Rotator Cuff Repair in Subjects Scheduled for a Repair Surgery.
Brief Title: InSpace™ System in Comparison to Best Repair of Massive Rotator Cuff Tear.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment target has not achieved due to very slow and low recruitment rate
Sponsor: OrthoSpace Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IS-CL-02-UK
Record Dates: First submitted 2014-08-03; First posted 2014-08-05 (Estimated); Last update posted 2020-06-05 (Actual); Status verified 2019-08

CONDITIONS: Full-thickness Rotator Cuff Tear
Keywords: Full-thickness/Massive Rotator Cuff Tear, Sub-acromial spacer

STUDY DESIGN:
Who Masked: Participant
Masking Description: The patient is blinded to the treatment type
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Best Repair of torn Rotator Cuff (Sham Comparator): Subjects will undergo surgical intervention (usually arthroscopy) to perform debridement, acromioplasty if deemed necessary, long head of biceps tenotomy, and at least partial repair.
  Interventions: Procedure: Best Repair of torn Rotator Cuff
- InSpace™ system (Active Comparator): Subjects will undergo surgical intervention (usually arthroscopy or mini invasive) of debridement, acromioplasty if deemed necessary with or without long head of biceps tenotomy, and placement of the InSpace™ system.
  Interventions: Device: InSpace™ system

INTERVENTIONS:
Procedure: Best Repair of torn Rotator Cuff
  Arms: Best Repair of torn Rotator Cuff
Device: InSpace™ system
  Arms: InSpace™ system

SUMMARY:
This is a post-marketing study to further assess the safety and effectiveness of the InSpace™ device implantation in comparison to surgical repair of full thickness Massive Rotator Cuff Tear .

DETAILED DESCRIPTION:
This is a post-marketing study to further assess the safety and effectiveness of the InSpace™ device implantation in comparison to surgical repair of full thickness Massive Rotator Cuff Tear .

The effectiveness will be assessed by comparing the shoulder outcome scores of each treatment arm ( ASES, Constant and Quick DASH) from pre-operation (baseline) up to 2 years post-operation, with respect to pain reduction, improvement of activity of daily living (ADL) and improvement of range of motion (ROM).

The safety will be asses by comparing the Adverse event rate between the treatment arms.

ELIGIBILITY:
Main Inclusion Criteria:

* Age 40 or older.
* Positive diagnostic imaging of the affected shoulder indicating full thickness Massive RCT involving more than one tendon.
* Persistent pain and functional disability of the affected shoulder for at least 3 months.

Main Exclusion Criteria :

* Known allergy to the balloon material (copolymer of PLA and -θ-caprolactone).
* Evidence of significant osteoarthritis or cartilage damage in the shoulder
* Evidence of gleno-humeral instability
* Previous surgery of the shoulder in the past 2 years, excluding diagnostic arthroscopy
* Evidence of major joint trauma, infection, or necrosis in the shoulder
* Partial-thickness tears of the rotator cuff

Ages: 40 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
The change in the Shoulder Score | baseline and 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Wigan and Leigh NHS Foundation Trust: Upper Limb & Trauma Surgery, Wigan, Hall Lane, Appley Bridge, United Kingdom